CLINICAL TRIAL: NCT04827875
Title: An Exploratory Study to Evaluate the Safety and Efficacy of Intradermal Administration of AIV001 Aqueous Suspension on Scar Formation and Keloid Recurrence Following Keloidectomy
Brief Title: Safety and Efficacy of AIV001 on Scar Formation and Keloid Recurrence Following Keloidectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AiViva BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AIV001-W02
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Keloid; Scar; Incision; Excision Margin
Keywords: Scar formation; Keloidectomy
MeSH Terms: conditions — Keloid; Cicatrix; Surgical Wound; Margins of Excision

STUDY DESIGN:
Intervention Model Description: Excisions of existing keloid scar, treatment of incisional area followed by evaluation of scar formation overtime.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AIV001 Treatment Dose 1 (Experimental): Intradermal, Dose 1
  Interventions: Drug: AIV001
- AIV001 Treatment Dose 2 (Experimental): Intradermal, Dose 2
  Interventions: Drug: AIV001

INTERVENTIONS:
Drug: AIV001 — Intradermal

SUMMARY:
To evaluate the saftye and effectiveness of AIV001 treatment on scar formation and/or keloid scar recurrence following keloidectomy.

DETAILED DESCRIPTION:
AIV001 (axitinib) has been formulated to provide focal disease-modifying therapy for patients undergoing surgical procedures where scar formation will occur. This was a multicenter, dose-escalation open label study to assess the safety and efficacy of AIV001 on scar formation and/or keloid recurrence following keloidectomy. This study design is an evaluation of surgical excision of keloid scar tissue followed by AIV001 intradermal injection. On Day 1, following keloidectomy, the incision area (devoid of keloid scar tissue) was sutured, creating an incision line. The incision line is the area of scar formation and assessment. This is a variable dose study defined by incision line length. The incision line length measurement defined each subject's AIV001 treatment based on the dose plan table in the protocol. Subjects received a minimum of 1 and up to 3 treatments, dependent on the protocol amendment implemented at the time of their participation and PI discretion based upon safety assessments. The excised tissue was sent to pathology for confirmation of keloid scar tissue. The treatment interval was Day 1 to Day 30 visits with observation visits on Days 60, 90, 183, and 365. A safety data review was conducted after the first 3 subjects in Cohort 1 completed the Day 30 visit. Assessment of local skin reactions (LSRs), wound healing, vitals, treatment-emergent adverse events (TEAEs) and pre-defined dose-limiting toxicities (DLTs) were reviewed to determine whether additional subjects were permitted to be enrolled. If safety was deemed acceptable, enrollment into Cohort 1 continued and Cohort 2 was open for enrollment. The same safety data review was conducted at Day 30 visit for the first 3 subjects enrolled in Cohort 2. The open-label study design allowed for adjustments to the dosing regimen (timing and frequency of dosing) based on review of each consecutive dosing cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male of female, aged 18 to 60, inclusive
* No clinically relevant abnormalities identified by a detailed medical history and vital signs
* Presence of one keloid scar, up to 2.2 cm length and up to 1.2 cm width, at least 1 year from formation, and located on trunk or arms
* Willing to undergo surgical excision of keloid
* No concurrent treatment of the study keloid or prior treatment within last 2 months

Exclusion Criteria:

* Prior keloidectomy of study keloid
* History of genetic disorder that predisposes to keloids (e.g., Ehlers-Danlos syndrome, Ullrich congenital muscular dystrophy, etc.)
* Corticosteroids (topical, injectable, inhalable, intranasal, or oral) within last two months (except as prescribed by physician for seasonal allergies)
* Clinically relevant cardiovascular, endocrine, hepatic, neurologic, renal, or other major systemic disease that could complicate execution of the protocol or interpretation of the study results
* History of thrombotic events, hemorrhagic events, and gastrointestinal perforation and fistula
* Subject has active collagen vascular disease or vasculitis, e.g., systemic lupus erythematosus, polyarthritis, dermatomyositis, systemic scleroderma or thrombotic thrombocytopenic purpura

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Adverse events | Approximately 365 days
  Incidence of adverse events

SECONDARY OUTCOMES:
Keloid recurrence | 365 days
  Number of subjects experiencing keloid recurrence within study duration
Modified Vancouver Scar Scale (mVSS) | Day 90 and Day 180
  Modified Vancouver Scar Scale (mVSS) includes four categories of scar quality (i.e., pliability (0-4), height (0-4), vascularity (0-3), and pigmentation (0-3)), with 0 representing normal body skin. The composite mVSS scar score (ranges 0-14) is the sum of the 4 category scores to represent the overall scar quality.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Skin Research Institute, Coral Gables, Florida
  - DermResearch DRI, Austin, Texas
  - J&S Studies, College Station, Texas